CLINICAL TRIAL: NCT04223817
Title: Contribution of 7.0 Tesla RMI in Screening of Osteoarticular Involvement and Vasculopathy of the Hands in Systemic Sclerosis
Brief Title: 7.0 Tesla Resonance Magnetic Imaging of the Hand in Systemic Sclerosis
Acronym: PREM'S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-A02760-57
Record Dates: First submitted 2019-12-30; First posted 2020-01-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Systemic Sclerosis (SSc); Magnetic Resonance Imaging (MRI)
Keywords: hand vascular involvement; hand osteoarticular involvement; magnetic resonnance imaging 7.0 tesla
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: SSc patients compared to control subjects without SSc matched on sex and age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7.0 Tesla MRI of both hands (Experimental): Single 7.0 Tesla MRI of both hands for all the SSc and control subjects
  Interventions: Device: 7.0 T RMI

INTERVENTIONS:
Device: 7.0 T RMI — Single 7.0 Tesla MRI of both hands in the same time

SUMMARY:
Systemic sclerosis (SSc) is a rare systemic autoimmune disease with specific osteoarticular pattern of unknown mechanism. Ischemic phenomenon have been suggested to participate to the osteoarticular involvement in SSc. To date, osteoarticular pattern and hand vascular involvement have been few studied in magnetic resonance imaging in SSc, and most often with low resolution RMI.

7 Tesla RMI allows high resolution for morphology examination, together with dynamic and functional vascular study and sodium articular concentration. Indeed, the aim of the study is to describe hand osteoarticular and vascular involvement in SSc, as well as sodium articular concentration. Clinico-biological association will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SSc:

  - ScS fulfilling ACR/EULAR 2013 classification criteria and followed in the department of internal medicine of Poitiers University Hospital, without clinical signs of digital arthrose
* Control subjects:

  - Hospitalized patients in the department of internal medicine of Poitiers University Hospital, without Raynaud's phenomenon, neither antecedent of inflammatory rheumatism and/or autoimmune disease, neither inflammatory articular symptoms during the previous month and no clinical signs of arthoses and/or arthritis at the inclusion in the study
* For both:

  * Age ≥ 18 years-old
  * Written informatory consent

Exclusion Criteria:

* Patients with SSc:

  - SSc associated with other define autoimmune disease (overlap syndrome)
* For both:

  * Absolute contraindication to 7.0 T RMI: pregnancy; ocular metallic foreign body ; cardiac pacemaker ; neurostimulator no compatible 7.0 T RMI ; cochlear implants; all electronic medical device implantedfor less than 6 weeks ; metallic heart valve ; old cranial vascular clips
  * Individuals with current health condition not allowing realization of the 7.0 T RMI in sufficient comfort conditions according to investigator appreciation (i.e. acute cardiac and/or respiratory failure, impossibility to maintain procubitus, bedridden individuals, claustrophobia)
  * Individuals under tutorship or guardianship
  * Individuals with reinforced protection: minors, judiciary or administrative decision
  * No affiliation to social insurance
  * Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Frequency of hand osteoarticular involvement in SSc and control subjects in 7.0 T RMI | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Frequency of type and localisation of hand osteoarticular abnormality (erosions, bone oedema, synovitis, tenosynovitis, intraarticular swoilling) in 7.0 T RMI in patients with SSc and control subjects

SECONDARY OUTCOMES:
Arterial pattern in the hand of SSc patients and control subjects in 7.0 T RMI | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Digital arteries count in both hand in 7.0 T RMI in SSc patients and control subjects
Arterial pattern in the hand of SSc patients and control subjects in 7.0 T RMI | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Lumen area of the selective section of the vessel (in mm2) in 7.0 T RMI in SSc patients and control subjects
Arterial pattern in the hand of SSc patients and control subjects in 7.0 T RMI | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Quality of arterial opacification in terms of percentage of digital artery that did not reach the first phalanx, in 7.0 T RMI in SSc patients and control subjects
Arterial pattern in the hand of SSc patients and control subjects in 7.0 T RMI | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Quality of venous return in terms of percentage of no visible venous return as far as the proximal phalanx in 7.0 T RMI in SSc patients and control subjects
Correlation between hand osteoarticular involvement in 7.0 T RMI and general and SSc-related factors, including hand vascular involvement, in SSc patients | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Proportion of hand osteoarticular abnormalities and : age (yrs) ; SSc duration (yrs) ; bone mass index ; modified Rodnan skin score (0-51) ; interlabial length (cm) ; arterial pattern in the hand in 7.0 T RMI ; proportions of female, active tabagism, SSc subtypes, SSc-related autoantibodies, antiphospholipid autoantibodies, immunosuppressant use, vasoactive drugs and SSc-related visceral involvement (Raynaud's phenomenon, digital tip ulcerations and/or gangrene and/or amputation, arterial pulmonary hypertension, interstitial lung disease, upper and/or lower digital tract involvement, renal crisis, arthritis, inflammatory myopathy, subcutaneous calcifications, telangiectasia) ; EUSTAR-Activity Index ; NT-proBNP level (ng/mL) ; troponin level (ng/mL) ; C reactive protein level (mg/L) ; proportion of capillaroscopic pattern (cutulo's classification) ; Raynaud's Condition Score ; patient's visual scale for Raynaud's phenomenon severity (1 to 10) ; SSc-HAQ ; "main de Cochin" score
Correlation between hand arterial involvement in 7.0 T RMI and general and SSc-related factors, including hand osteoarticular involvement, in SSc patients | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Proportion of hand hand arterial abnormalities and : age (yrs) ; SSc duration (yrs) ; bone mass index ; modified Rodnan skin score (0-51) ; interlabial length (cm) ; hand osteoarticular abnormalities in 7.0 T RMI ; proportions of female, active tabagism, SSc subtypes, SSc-related autoantibodies, antiphospholipid autoantibodies, immunosuppressant use, vasoactive drugs and SSc-related visceral involvement (Raynaud's phenomenon, digital tip ulcerations and/or gangrene and/or amputation, arterial pulmonary hypertension, interstitial lung disease, upper and/or lower digital tract involvement, renal crisis, arthritis, inflammatory myopathy, subcutaneous calcifications, telangiectasia) ; EUSTAR-Activity Index ; NT-proBNP level (ng/mL) ; troponin level (ng/mL) ; C reactive protein level (mg/L) ; proportion of capillaroscopic pattern (cutulo's classification) ; Raynaud's Condition Score ; patient's visual scale for Raynaud's phenomenon severity (1 to 10) ; SSc-HAQ ; "main de Cochin" score
Sodium articular concentration in the hand in 7.0 T RMI in SSc patients and control subjects | 7 days maximum (delay between realization of the RMI and its final interpretation)
  Mean values of sodium articular concentration in the hands of SSc patients of control subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided